CLINICAL TRIAL: NCT03538509
Title: Percutaneous Coronary Intervention in Patients witH OrthotoPic hEart Transplantation: the PCI-HOPE a Multicenter Study
Acronym: PCI-HOPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fabrizio D'Ascenzo (Other)
Collaborators: University of Zurich (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); University of Padova (Other); University of Bologna (Other); Hospital Clinic of Barcelona (Other); University of Roma La Sapienza (Other)
Responsible Party: Sponsor-Investigator, Fabrizio D'Ascenzo, Medical Doctor, A.O.U. Città della Salute e della Scienza
Organization: A.O.U. Città della Salute e della Scienza (Other)
Other Study IDs: PCI-HOPE
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Heart Transplant Failure and Rejection; Coronary Artery Disease
MeSH Terms: conditions — Rejection, Psychology; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PCI and implantation drug eluting stent or bare metal stent — Percutaneous Coronary Angioplasty

SUMMARY:
This is a retrospective, multicenter, study including patients undergone to one or more percutaneous revascularization after OHT. The rate of restenosis, the kind of percutaneous revascularization, the feature of coronary disease and the medical therapy for positive vessel remodeling will be evaluated.

DETAILED DESCRIPTION:
Actual standard of care. Orthotopic heart transplantation (OHT) represents the optimal solution for the cure of end-stage heart failure, but it is burdened by numerous comorbidity. The main cause of morbidity and mortality in these patients is related to Transplant coronary artery disease (TCAD), that affects at least fifth percent of transplanted at five years of transplantation. TCAD is a purely immunological phenomen, emphasized by non-immunological factors, favoring oxidative stress, like dyslipidemia, smoking, hypertension, diabetes.(1-3) Many anatomic-pathological studies showed cellular infiltration with predominance of T-cell, mainly in the neointima and in adventizia. TCAD often resulted without angor because of denervation of the heart after transplantation (4-6). The managment and the treatment of TCAD are somewhat complex, because of accelerated vasal infiltration. Furthermore in multivessel disease a surgery revascularisation presented an elevated surgery risk.

Limits and complications of actual standard of care. In the first era of angioplasty percutaneous therapy was considered like palliation in this kind of coronary lesions , but with the beginning of BMS and DES era the outcomes of these patients considerably improved. However TCAD's lesions showed a rate of restenosis greater than classic atherosclerotic plaques(7). There is also a disagreement of results between implantation of DES or BMS, because some studies showed a superiority of the DES group, others didn't show any significant difference(8-9).

Potential improvements of standard of care. In this retrospective study an interesting point of research would be point out if the risk of restenosis was reduced with a particular kind of medicated stent for local effect of polymers, currently used. The general pharmacological effect of sirolimus was known like inhibitor of cell-T proliferation and then it could reduce vessel cellular infiltration, acting as a local immunosuppressant(10-12).

For this argument evidence is discordant, although the problem is getting relevant due to the prolonged survival of these patients and the augmented number of transplantation. These patients are often young and have an elevated general risk for iatrogenic immunosuppressed state. Therefore with this retrospective study we propose to understand the physio-pathological mechanisms of TCAD and also what actual therapy results the best .

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergone percutaneous revascularization, both with symptomatic CAD and asymptomatic, with one or more coronary vessel disease, will be enrolled.

Exclusion Criteria:

1. Infective endocarditis;
2. Life expectancy less than 1 year for non-cardiovascular causes;
3. Recent cerebrovascular accident (<6 months);
4. Inability to express informed consent;

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Evaluation incidence, prognostic factors and outcomes of percutaneous theraphy in patients with Transplant Coronary Artery Disease (TCAD)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of restenosis | 18 years
  observation rate of restenosis post-PCI

SECONDARY OUTCOMES:
MACE | 18 years
  Number of Cardiovascular events
Rate of TCAD | 18 years
  Number of CAD in transplant recipients

CONTACTS AND LOCATIONS:
Locations (1):
- Citta della Salute, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmer RJ, Lee MS. Transplant coronary artery disease. JACC Cardiovasc Interv. 2010 Apr;3(4):367-77. doi: 10.1016/j.jcin.2010.02.007. PMID 20398862